CLINICAL TRIAL: NCT06245967
Title: Frequency Specific Microcurrent Therapy for Mild Traumatic Brain injury-a Single Center Double-blind Randomized Sham-controlled Trail
Brief Title: Frequency Specific Microcurrent Therapy for Mild Traumatic Brain Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMUH112-REC3-176
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Trauma, Head; Headaches Posttraumatic; Dizziness; Brain Concussion; Frequency Specific Microcurrent Therapy
Keywords: Frequency specific microcurrent therapy; Concussion; Traumatic brain injury
MeSH Terms: conditions — Craniocerebral Trauma; Post-Traumatic Headache; Dizziness; Brain Concussion; Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): True FSM (Concussion protocol) with symptom management medication
  Interventions: Device: Frequency specific microcurrent therapy
- Sham-control (Sham Comparator): Sham FSM (no protocol) with symptom management medication
  Interventions: Device: Sham Frequency specific microcurrent therapy

INTERVENTIONS:
Device: Frequency specific microcurrent therapy — Concussion protocol
  Arms: Experimental
Device: Sham Frequency specific microcurrent therapy — Shan concussion protocol
  Arms: Sham-control

SUMMARY:
Patients with mild traumatic brain injury (mTBI) may experience spontaneous recovery within 7-10 days, but some continue to exhibit symptoms such as headache, dizziness, vertigo, poor concentration, and cognitive dysfunction. Effective treatments for these symptoms are currently lacking. Frequency Specific Microcurrent(FSM) has received approval from the U.S. FDA for use in neuroinflammatory conditions. Our study aims to evaluate the efficacy of FSM by using FSM device ,IS02LCDs Stimulator (Ru Yi Health ltd. Co,Taiwan R.O.C), on symptom improvement in 52 patients with mild TBI

DETAILED DESCRIPTION:
This study is a single center double-blind randomized sham-controlled trail.We aims to recruit 52 mild traumatic brain injury participants with symptoms for more than 10 days.Clinical assessments include Post-Concussion Symptom Scale (PCSS) scores, and the amount of medication used for symptom management. These 52 participants will be 1:1 randomly allocated into two groups (1) sham FSM with symptom management medication and (2) True FSM with symptom management medication. The treatment period will last two weeks, with a total of six therapy sessions. Following treatment, a four-week observation period will be conducted. The primary outcome measurement will be changes in the Post-Concussion Symptom Scale (PCSS) scores, recorded at baseline, after the third treatment session, at the end of treatment, and at the end of the observation period. Secondary outcome measures will include the amount of medication used for symptom management. The safety evaluated index is the adverse event rate for two groups. These assessments aim to evaluate the therapeutic benefits of FSM for mild traumatic brain injury.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20 and 65, inclusive, for both males and females.
2. History of traumatic brain injury with a loss of consciousness lasting less than 30 minutes, initial Glasgow Coma Scale (GCS) score ranging from 13 to 15.
3. Presence of persistent post-concussion symptoms starting from the day of injury and lasting for more than ten days.
4. Complete consciousness or decision-making capacity at the time of enrollment.
5. Brain imaging through CT or MRI indicating the absence of significant midline shift, no evident damage to the brainstem (excluding the pyramidal tract), or thalamus. Each brain lobe lesion should not exceed 30% of the respective cerebral hemisphere.

Exclusion Criteria:

1. Individuals below 20 years or above 65 years of age, regardless of gender.
2. History of traumatic brain injury with a loss of consciousness exceeding 30 minutes, initial Glasgow Coma Scale (GCS) score less than 13.
3. Not a first-time occurrence of traumatic brain injury.
4. Brain imaging through CT or MRI revealing significant midline shift, evident damage to the brainstem or thalamus, with each brain lobe lesion exceeding 30% of the respective cerebral hemisphere.
5. Presence of comorbidities such as cancer, depression.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Post-Concussion Symptom Scale (PCSS) scores | 1.5 month
  The Post-Concussion Symptom Scale (PCSS) is used to assess the number and intensity of symptoms after a concussion/mild traumatic brain injury.

SECONDARY OUTCOMES:
the amount of medication used for symptom management | 1.5 month
  the amount of medication used for symptom management

CONTACTS AND LOCATIONS:
Overall Officials: I HAN Hsiao, Principal Investigator — China Medical University Hospital

IPD SHARING:
Plan to Share IPD: No